CLINICAL TRIAL: NCT06697665
Title: An Exploratory Clinical Study to Evaluate the Safety, Tolerability, Immune Response and Preliminary Efficacy of LM103 Injection in Combination With PD-1 in Patients With Advanced Solid Tumours
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Suzhou BlueHorse Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LM-CM-TIL
Record Dates: First submitted 2024-11-15; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Solid Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant Group (Experimental): Treatment includes LM103 injection and PD-1
  Interventions: Biological: LM103

INTERVENTIONS:
Biological: LM103 — Patients were treated with PD-1, cyclophosphamide and fludarabine, LM103 and IL-2 treatment.

SUMMARY:
This is an exploratory clinical study evaluating the safety, tolerability, immune response and preliminary efficacy of LM103 Injection in combination with PD-1 in patients with advanced solid tumours. The research treatment includes LM103 injection, IL-2 therapy, PD-1 therapy,fludarabine and cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

1. The expected survival time is not less than 3 months.
2. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0-1.
3. Patients with advanced solid tumors confirmed by histology or cytology: advanced Melanoma, cervical cancer/ovarian cancer, head and neck squamous cell cancer, non-small cell lung cancer, esophageal cancer and other solid tumors that have failed standard treatment regimens, cannot tolerate standard treatment, refuse or do not have standard treatment regimens available.
4. The patient has lesions that can be used for surgical resection (>1.5 cm3) or biopsy puncture (no less than 6 lesions) for LM103 manufacturing.
5. At least one measurable lesion as the target lesion after collecting tumor tissue from the patient (RECIST v1.1 criteria).
6. Laboratory tests results during the screening period indicate that the subjects have sufficient organ function.

Exclusion Criteria:

1. Have a medical history of other malignant tumors other than the disease under study in the past 5 years, except for malignant tumors that can be expected to recover after treatment (including but not limited to thyroid cancer, cervical Carcinoma in situ, basal or squamous cell skin cancer or Ductal carcinoma in situ of the breast treated by radical surgery).
2. LM103 received systematic therapy of antineoplastic drugs (including chemotherapy, small molecule targeted drug therapy, Hormone replacement therapy, etc.), or local antineoplastic therapy (such as radiotherapy, palliative radiotherapy for bone metastases>2 weeks before the start of the study and intracranial stereotactic radiotherapy or resection of a single brain metastasis>3 weeks before the start of the study were acceptable) within 4 weeks before LM103 infusion; Or received clinical investigational drugs or equipment treatment.
3. Adverse reactions caused by previous treatment have not recovered to CTCAE (version 5.0) level 1 or below (excluding hair loss and neurotoxicity, which have been determined by the researchers to be irreparable and level 2 hypothyroidism for a long time).
4. Previously received allogeneic hematopoietic stem cell transplantation or solid organ transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AE), Serious adverse event (SAE) and immune related adverse events (irAE) | through study completion, an average of 1 year estimate
  Incidence and severity of AE, SAE and irAE; Abnormal changes in laboratory and other tests with clinical significance.

SECONDARY OUTCOMES:
Objective response rate (ORR) | through study completion, an average of 1 year estimate
  The Objective Response Rate (ORR) was defined as the percentage of participants who achieved a best overall response of confirmed Complete Response (CR) or Partial Response (PR), assessed by investigator assessment based on RECIST version 1.1.
Duration of response (DOR) | through study completion, an average of 1 year estimate
  Duration of Response (DOR) was defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first objective documentation of progressive disease (PD) or death due to any cause.
Disease control rate (DCR) | through study completion, an average of 1 year estimate
  Disease control rate (DCR) was defined as the percentage of participants with a best overall response of CR, PR or SD as defined by RECIST version 1.1.
Time to response (TTR) | through study completion, an average of 1 year estimate
  Time to progression (TTP) is defined as the interval between the date of randomization and the earliest date of progression of disease (PD) or death due to the solid tomor.
Time to disease progression (TTP) | through study completion, an average of 1 year estimate
  Time to progression (TTP) is defined as the interval between the date of randomization and the earliest date of progression of disease (PD) or death due to the solid tomor.
Progression free survival (PFS) | through study completion, an average of 1 year estimate
  Progression-free survival (PFS) was defined as the time from the date of enrollment to the earlier of the dates of the first objective documentation of disease progression (as per RECIST version 1.1) or death due to any cause.
Overall survival (OS) | through study completion, an average of 1 year estimate
  OS was defined as the time from first dose to date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Beichen Hospital, China, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided